CLINICAL TRIAL: NCT06045091
Title: A Early Phase 1 Clinical Trial to Evaluate the Safety and Efficacy of Human BCMA Targeted CAR-NK Cells Injection for Subjects With Relapsed/Refractory Multiple Myeloma or Plasma Cell Leukemia
Brief Title: To Evaluate the Safety and Efficacy of Human BCMA Targeted CAR-NK Cells Injection for Subjects With R/R MM or PCL
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRAIN01-MM04-POC
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma; Plasma Cell Leukemia
Keywords: BCMA; CAR-NK; Multiple Myeloma; Plasma Cell Leukemia; Relapsed /Refractory
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human BCMA Targeted CAR-NK Cells Injection (Experimental): Two doses on Day 0 and Day 7. 1.5×10^8 CAR+NK cells/dose, 3.0×10^8 CAR+NK cells/dose or 6.0×10^8 CAR+NK cells/dose
  Interventions: Drug: Human BCMA targeted CAR-NK cells injection

INTERVENTIONS:
Drug: Human BCMA targeted CAR-NK cells injection — Allogenic genetically modified anti-BCMA CAR transduced NK cells
  Other Names: BCMA CAR-NK

SUMMARY:
This study is a single-arm, open-label, dose-escalation trial to explore the safety, tolerability and pharmacokinetic/pharmacodynamics characteristics of human BCMA targeted CAR-NK Cells injection, and to preliminarily observe the efficacy of the trial drug in patients with relapsed/refractory multiple myeloma or plasma cell leukemia.

DETAILED DESCRIPTION:
Subjects with relapsed/refractory multiple myeloma or plasma cell leukemia can participate if all eligibility criteria are met. Tests required to determine eligibility including disease assessments, a physical exam, Electrocardiograph, Computed tomography (CT)/Magnetic Resonance Imaging (MRI)/Positron Emission Tomography (PET), liver/renal function tests, complete blood count with differential and complete metabolic profile and etc. Subjects will receive preconditioning chemotherapy prior to the first infusion of human BCMA targeted CAR-NK Cells injection. After the infusion, subjects will be followed for adverse events, pharmacokinetic/pharmacodynamics characteristics, efficacy of human BCMA targeted CAR-NK cells. Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:Subjects must meet all of the following criteria to be enrolled:

* Subjects volunteer to participate in clinical trials, understand and sign the informed consent document, be willing to complete all the trial procedures;
* 18 years and older, Male and female;
* Expected survival > 12 weeks;
* Documented evidence of multiple myeloma at diagnosis as defined by IMWG updated criteria (2014), or plasma cell leukemia at diagnosis as defined by Diagnosis and therapeutic criteria of hematologic disease (4th edition);
* One of the following indicators is satisfied:

  1. Serum M protein: IgG M protein ≥5 g/L; or IgA M protein ≥5 g/L; or IgD M protein and IgD >ULN;
  2. Urine M protein ≥200 mg/24h;
  3. Affected serum free light chain ≥100 mg/L and Serum free light chain ratio is abnormal;
  4. Clonal bone marrow plasma cells ≥10 % for non-secretory myeloma;
* Patients with relapsed/refractory multiple myeloma or plasma cell leukemia, satisfying:

  1. Patients have received at least 3 prior MM or PCL treatment regimens containing at least one proteasome inhibitor and one immunomodulatory;
  2. Progress is documented within 60 days of the most recent anti-tumor treatment, or efficacy assessment does not reach minimal response(MR) or above;
* Liver, kidney and cardiopulmonary functions meet the following requirements:

  1. Creatinine clearance rate (estimated by CockcroftGault formula) ≥30mL/min;
  2. Left ventricular ejection fraction > 50%;
  3. Baseline peripheral oxygen saturation > 95%;
  4. Total bilirubin≤ 2×ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN;
* Blood routine examination satisfying hemoglobin≥60 g/L, neutrophils≥ 1.0×10^9/L, and platelets≥30×10^9/L, can complete this trial according to the judgement of investigators.

Exclusion Criteria:Any one of the following conditions cannot be selected as a subject：

* Accompanied by other uncontrolled malignancies;
* Subjects with positive Hepatitis B surface antigen(HBsAg) or Hepatitis B core antibody (HBcAb) and hepatitis B virus (HBV) DNA titers higher than the lower limit of the normal range of the investigative site; Hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; Human Immunodeficiency Viral (HIV) antibody positive; syphilis primary screening antibody positive;
* Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia, liver, kidney, or metabolic disease;
* Subjects who are considered unsuitable to participate in this trial by the investigator.
* Pregnant or lactating woman, and female subject who plans to have a pregnancy within 1 year after cell transfusion, or male subject whose partner plans to have a pregnancy within 1 year after cell transfusion;
* Received CAR-NK treatment or other gene therapies before enrollment;
* Subjects who have a disease that affects the signing of written informed consent or who are unable to comply with research procedures; or who are unwilling or unable to comply with research requirements;
* Subjects who have had severe immediate hypersensitivity reactions to any drugs used in this research;
* Active or uncontrollable infection requiring systemic therapy within 14 days prior to enrollment;
* In the past two years, the terminal organ was damaged due to autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus), or the systemic use of immunosuppressive or other systemic disease control drugs was required;
* Patients with symptoms of central nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) | 28 days post infusion
  Safety Indicators

SECONDARY OUTCOMES:
Pharmacokinetics parameters - the highest concentration of human BCMA targeted CAR-NK cells amplified in peripheral blood and bone marrow after infusion | 2 years post infusion
  Effectiveness Metrics
Pharmacokinetics parameters - the time to reach the highest concentration of human BCMA targeted CAR-NK cells amplified in peripheral blood and bone marrow after infusion | 2 years post infusion
  Effectiveness Metrics
Pharmacokinetics parameters - the 28-day area under the curve of human BCMA targeted CAR-NK cells amplified in peripheral blood and bone marrow after infusion | 2 years post infusion
  Effectiveness Metrics
Pharmacodynamics characteristics - the detection values of CRP, IL-6, IL-15, Granzyme B cytokines in peripheral blood | 2 years post infusion
  Effectiveness Metrics
Pharmacodynamics characteristics - the detection values of monoclonal plasma cell in bone marrow | 2 years post infusion
  Effectiveness Metrics
Overall response rate (ORR, include PR, VGPR, CR and sCR) after administration | 3 months post infusion
  Effectiveness Metrics
Percentage of subjects with negative minimal residual disease (MRD) | 2 years post infusion
  Effectiveness Metrics
Duration of subjects with negative minimal residual disease (MRD) | 2 years post infusion
  Effectiveness Metrics
Number of subjects with adverse events | 2 years post infusion
  Safety Metrics
Change from baseline in perform status as measured by Easten Cooperative Oncology Group (ECOG) score | Safety Metrics
  2 years post infusion
The occurrence rate of adverse events grade≥3 assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. | 2 years post infusion
  Safety Metrics
Change in body weight over time after infusion | 2 years post infusion
  Safety Metrics
Duration of remission (DOR) after administration | 2 years post infusion
  Effectiveness Metrics
Overall Survival (OS) after administration | 2 years post infusion
  Effectiveness Metrics

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, Doctor, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No